CLINICAL TRIAL: NCT05079854
Title: Use Of Intracameral Moxifloxacin For Prophylaxis Of Open Globe Endophthalmitis
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Federal University of São Paulo (Other)
Responsible Party: Principal Investigator, Mauricio Maia, Clinical Professor, Federal University of São Paulo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: TOP_VIGAMOX
Record Dates: First submitted 2021-10-03; First posted 2021-10-15 (Actual); Last update posted 2021-11-10 (Actual); Status verified 2021-11

CONDITIONS: Endophthalmitis; Trauma, Corneal
MeSH Terms: conditions — Endophthalmitis; Corneal Injuries | interventions — Intracameral Injection

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- INTRACAMERAL MOXIFLOXACIN (Active Comparator): After the surgery, the antibiotic is intracameral administered, Moxifloxacin 0.5% 0.1mL.
  Interventions: Drug: Intraocular Instillation Solution
- TOPICAL MOXIFLOXACIN (Active Comparator): After the surgery, the antibiotic is topical administered, Moxifloxacin 0.5% 0.1mL.
  Interventions: Drug: Moxifloxacin Ophthalmic

INTERVENTIONS:
Drug: Intraocular Instillation Solution — Intracameral Moxifloxacin 0.5%
  Other Names: Intracameral
  Arms: INTRACAMERAL MOXIFLOXACIN
Drug: Moxifloxacin Ophthalmic — Topical Moxifloxacin 0.5%
  Arms: TOPICAL MOXIFLOXACIN

SUMMARY:
Endophthalmitis is a severe inflammatory eye condition with profound impairment of vision, which can lead to irreversible visual loss and requires immediate treatment.

There is no way to completely prevent endophthalmitis, however, through prophylactic methods, it is possible to reduce its incidence. Currently, the only technique that has reached category II of evidence in reducing the risks of endophthalmitis is the use of 5% povidone-iodine eye drops, moments before surgery. In 2007, the European Society of Cataract and Refractive Surgery (ESCRS) released a large multicenter randomized clinical trial, with data on the reduction in the rates of endophthalmitis, using the intracameral antibiotic therapy technique of perioperative cefuroxime. However, much is discussed about the risks related to the technique, such as dilutional errors, contamination, anaphylaxis and cost-effectiveness, which still makes the conduct debatable.

The study evaluates the use of intracameral Moxifloxacin 0.5% (Vigamox®) as prophylaxis in cases of endophthalmitis after open ocular trauma;

ELIGIBILITY:
Inclusion Criteria:

* open globe trauma

Exclusion Criteria:

* endophthalmitis at the beginning

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2023-11-01 (Estimated)

PRIMARY OUTCOMES:
Endophthalmitis | 90 days
  Evaluate the incidence of Endophthalmitis

CONTACTS AND LOCATIONS:
Locations (1):
- Dept of Ophthalmology - UNIFESP/Hospital São Paulo, São Paulo, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol